CLINICAL TRIAL: NCT07123324
Title: Prospective Multicenter Observational Study of the Management and Prognosis of Severe Acute Kidney Injury (AKI) in Nephrology Units: The French AKI Registry (FAKIR)
Brief Title: French AKI Registry (FAKIR): A Multicenter Study on the In-Hospital Management and Outcomes of Severe Acute Kidney Injury in Nephrology Units
Acronym: FAKIR
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9876
Record Dates: First submitted 2025-08-07; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Acute Kidney Injury; Kidney Failure Chronic; Cardiorenal Syndrome; Renal Replacement Therapies; Hospitalizations
Keywords: Kidney injury; Renal function recovery; Dialysis initiation; Kidney biopsy; Cardiovascular complications; Nephrology care; Renal prognosis; Renal cohort; Kidney follow-up; Kidney disease progression
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency, Chronic; Cardio-Renal Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AKI KDIGO 2-3 Nephrology Patients: This cohort includes adult patients (≥18 years old) hospitalized in nephrology wards (including conventional units and nephrology intensive care) for acute kidney injury (AKI) classified as KDIGO stage 2 or 3 at admission. Patients with AKI acquired outside nephrology or limited to stage 1 are excluded. Clinical data will be collected during hospitalization and follow-up visits at 3, 6, and 12 months to assess renal recovery, progression to chronic kidney disease, major cardiovascular events, and mortality. This group represents real-life management of severe AKI in nephrology units across multiple centers.

SUMMARY:
Acute Kidney Injury (AKI) is a common and serious condition in hospitalized patients, especially when it reaches stages 2 or 3 according to the KDIGO classification. These severe forms are associated with high mortality, a risk of progression to chronic kidney disease (CKD), and frequent cardiovascular complications. However, current data on how nephrologists manage these patients during hospitalization-and how these practices influence long-term outcomes-are limited and heterogeneous.

The FAKIR study (French AKI Registry) is a prospective, multicenter, non-interventional observational study designed to describe the clinical management of patients admitted to nephrology departments for AKI stage 2 or 3 and to assess their renal and cardiovascular outcomes up to one year. The study hypothesizes that better characterization of in-hospital practices and patient trajectories will help identify predictors of renal recovery, progression to end-stage renal disease, and major cardiovascular events.

Patients will be followed during hospitalization and at 3, 6, and 12 months to assess renal function, mortality, cardiovascular events, and rehospitalizations. This registry aims to provide real-life, multicenter data to support future guidelines and the development of structured post-AKI care pathways.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at admission
* Hospitalized in a nephrology ward (standard or intensive nephrology care unit)
* Diagnosis of acute kidney injury (AKI) stage 2 or 3 according to KDIGO criteria at the time of admission
* Availability of follow-up data at 3 months (clinical or laboratory)

Exclusion Criteria:

* AKI stage 1 only
* AKI acquired outside the nephrology department without subsequent transfer to nephrology
* Hospitalized for another reason without documented AKI stage 2 or 3
* Refusal or opposition to data reuse for research purposes
* Under legal protection (guardianship or trusteeship) without a representative to provide non-opposition
* Incomplete medical records preventing collection of required baseline data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients (≥18 years) hospitalized in nephrology departments across multiple French university hospitals for acute kidney injury (AKI) stage 2 or 3. Patients are identified prospectively at the time of admission to nephrology units, either directly or via transfer from emergency or other hospital departments. Only patients with confirmed KDIGO stage 2 or 3 AKI at admission are included. Data are collected during hospitalization and up to 12 months post-discharge to assess renal and cardiovascular outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Complete Renal Recovery at 3 Months After Hospitalization for AKI KDIGO Stage 2 or 3 | Assessed at 3 months (±30 days) after admission for AKI in nephrology ward
  Renal recovery is defined as a return of serum creatinine to ≤125% of the patient's baseline (pre-AKI) value, estimated using the CKD-EPI formula. Creatinine values are collected from medical records or follow-up labs performed at 3 months post-discharge. This outcome reflects the extent of renal function recovery following hospitalization for severe AKI and helps identify prognostic factors associated with favorable evolution.

SECONDARY OUTCOMES:
All-Cause Mortality at 12 Months After Hospitalization for AKI KDIGO Stage 2 or 3 | Assessed at 12 months post-admission (±30 days)
  All-cause mortality is defined as the proportion of patients who die from any cause within 12 months following their admission for AKI KDIGO stage 2 or 3. Vital status is obtained from hospital records, follow-up contact, or national registries. This outcome will allow assessment of medium-term prognosis and identification of clinical factors associated with mortality in patients with severe AKI managed in nephrology units.
Incidence of Major Adverse Cardiovascular Events (MACE) at 12 Months | Assessed throughout the 12-month follow-up period
  MACE includes non-fatal myocardial infarction, non-fatal stroke, hospitalization for acute heart failure, and cardiovascular death. Events will be identified from medical records, discharge summaries, and follow-up contacts. This outcome will assess the cardiovascular burden among patients with severe AKI managed in nephrology settings, and help determine the link between in-hospital management strategies and long-term cardiovascular risk.
Progression to End-Stage Renal Disease (ESRD) at 12 Months | Assessed at 12 months post-AKI hospitalization
  ESRD is defined as the initiation of chronic renal replacement therapy (dialysis or kidney transplantation) or a sustained eGFR <15 mL/min/1.73m². Data are collected through follow-up visits, patient contact, or hospital records. This measure evaluates long-term renal outcomes and identifies risk factors for irreversible kidney failure following AKI KDIGO stage 2 or 3.

IPD SHARING:
Plan to Share IPD: Undecided